CLINICAL TRIAL: NCT04739033
Title: Lifestyle Online Intervention On Eating Behaviour and Body Mass Index On Obese Hypertensive Adults
Brief Title: Lifestyle Online Intervention On EB and BMI On Obese Hypertensive Adults
Acronym: LOIEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor of the Deparment of Biomedical Sciences, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCH-86
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension; Obesity; Internet; Exercise; Nutrition; Eating Behaviour
MeSH Terms: conditions — Hypertension; Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.
  The self-applied online program will comprise a three months behavioural intervention composed by 9 modules seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.
  Interventions: Behavioral: VIVIR MEJOR EXPERIMENTAL
- Control Group (Active Comparator): The control group will receive the same webbased lifestyle intervention (exercise and nutritional education), but in this case supported by audiovisual instructions given by a doctor outside the patient.
  Interventions: Behavioral: VIVIR MEJOR EXPERIMENTAL

INTERVENTIONS:
Behavioral: VIVIR MEJOR EXPERIMENTAL — This group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.
  The self-applied online program will comprise a three months behavioural intervention composed by 9 modules seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.

SUMMARY:
This study aims to analyze the effects of a online program focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on obese or overweight adults with hypertension. Participants will be recruited from a hypertension unit of a public hospital. These patients will be randomized allocated into two interventional groups: experimental group will receive audiovisual instructions from their hypertension specialist doctor, and the control group from a doctor outside the patient. Assessment will include: body composition (BMI), blood pressure, and eating behaviour.

DETAILED DESCRIPTION:
Hypertension incidence and overweight or obesity related, constitute a worrying public health problem nowadays. Evidence indicates that, despite the existence of several factors involved in their etiology, diet and physical activity play a particularly important role in the treatment and prevention of obesity and associated disorders. However, interventions for the treatment of obesity encounter some environmental and personal barriers, specifically problems or deficits in motivation. These barriers sometimes make it difficult to implement intervention strategies. In this sense, there is an important agreement about the need to generate alternatives and strategies which promote intrinsic motivation, self-regulation and self-efficacy as fundamental variables which have a direct relationship with the adherence and success of obesity treatments. To achieve this, Information and Communication Technologies (ICTs) are a very promising alternative, as they can provide personalised feedback and can be flexibly adapted to each user. In addition, ICTs also present other important advantages, especially their excellent cost-benefit ratio, and the possibility of increasing the efficiency of the interventions, since they allow to reach a greater number of users at a lower cost.

Therefore, this study aims to analyze the effects of a 3 months duration self-applied online program, composed of 9 modules focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on obese or overweight adults with hypertension. Participants will be recruited from a hypertension unit of a public hospital. These patients will be randomized allocated into two interventional groups: experimental group will receive audiovisual instructions from their hypertension specialist doctor, and the control group from a doctor outside the patient. Assessment will include: body composition (BMI), blood pressure, and eating behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Overweight or obesity (25 ≤ BMI ≤ 35 kg/m2)
* Aged between 18-75 years
* Being a participant of the program 5 years ago

Exclusion Criteria:

* Not having access to the Internet or lack of information about it.
* Treatment with more than 3 antihypertensive drugs.
* Meet the criteria of the DSM-IV-TR of a Food Disorder.
* Presenting some type of severe psychiatric disorder.
* Disability that prevents or hinders physical exercise.
* Receiving some treatment for weight loss.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Eating Behaviour, as measured with the DEBQ (Dutch Eating Behaviour Questionnaire). | 3 months
  The Dutch Eating Behaviour Questionnaire has 33 items, 13 of which refer to the emotional eating scale (eg, 'Desire to eat when irritated') and 10 of which refer to the external (eg, 'Eating when you feel lonely') and restrictive (eg, 'Difficult to resist delicious food') scales. The items can be rated on a five-point Likert-type scale, with a score of 1 indicating 'never' and 5 indicating 'very often (range 33-165). The lower the scores are, the lower the problematic eating behaviours are.

SECONDARY OUTCOMES:
BMI | 3 months
  Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, Principal Investigator — Cardenal Herrera University
Locations (1):
- Juan Francisco Lisón Párraga, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lison JF, Palomar G, Mensorio MS, Banos RM, Cebolla-Marti A, Botella C, Benavent-Caballer V, Rodilla E. Impact of a Web-Based Exercise and Nutritional Education Intervention in Patients Who Are Obese With Hypertension: Randomized Wait-List Controlled Trial. J Med Internet Res. 2020 Apr 14;22(4):e14196. doi: 10.2196/14196. PMID 32286232